CLINICAL TRIAL: NCT05642026
Title: The Efficacy of Continuous Intercostal Nerve Blocks in the Treatment of Patients With Multiple Rib Fractures
Brief Title: INTERCOSTAL NERVE BLOCK: Efficacy of CINB for Patients With Multiple Rib Fractures
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zachary Warriner (Other)
Responsible Party: Sponsor-Investigator, Zachary Warriner, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SURMI-22-INTERCOSTAL-NB
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Rib Fractures
Keywords: intercostal; nerve block; opioid; non steroidal; inpatient; outpatient; catheter; anesthetic; epidural
MeSH Terms: conditions — Rib Fractures | interventions — Ropivacaine; Anti-Inflammatory Agents, Non-Steroidal; Analgesics, Opioid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- continuous intercostal nerve block (CINB) (Experimental): patients admitted to the adult trauma service with rib fractures who are receiving CINB
  Interventions: Drug: Ropivacaine; Drug: Non steroidal anti-inflammatory drug and opioids
- standard medical care (Active Comparator): patients admitted to the adult trauma service with rib fractures who are receiving standard medical care
  Interventions: Drug: Non steroidal anti-inflammatory drug and opioids

INTERVENTIONS:
Drug: Ropivacaine — Patients in this group will receive CINB (continuous local intercostal infusion of 0.2% Ropivacaine). A single catheter will be placed for short segment involvement and two catheters will be placed in series for longer segments of involvement. If necessary and as part of standard of care, CINB treatment will continue after patient discharge. The administration of CINB therapy will continue in the same manner as inpatient therapy.
  Other Names: Naropin
  Arms: continuous intercostal nerve block (CINB)
Drug: Non steroidal anti-inflammatory drug and opioids — Patients in this group receive nonsteroidal and opioid pain medications (intravenous/oral inpatient and oral outpatient) per standard of care.

SUMMARY:
This is a prospective, randomized, non-blinded study comparing CINB plus medical therapy versus standard medical care (non-steroidals and opioids intravenous/oral inpatient and oral outpatient) alone for patients with multiple rib fractures. The objective of this study is to analyze the effect of continuous intercostal nerve block (CINB) in the treatment of patients admitted to the adult trauma service with rib fractures. The effectiveness of CINB as adjunctive treatment will be compared to standard medical therapy involving nonsteroidal and intravenous/oral opioid medications.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be at least 18 years old
* Subjects will have 2 or more identified rib fractures
* Subjects will be willing to provide informed consent for procedure
* Subjects will be identified as appropriate for initiation of continuous nerve block therapy for treatment of rib fracture associated pain.

Exclusion Criteria:

* Documented allergy to study medication
* Epidural catheter use
* Prisoners
* Refusal of CINB therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | 7 days
  time from randomization until the time of discharge

SECONDARY OUTCOMES:
Patient daily pain scores | 7 days
  Pain will be assessed using a 10-Point Numerical Pain Scale (as part of standard of care) every day while patient is hospitalized and 2 days following discharge at follow contact. Scores range from 0-10; higher scores indicated higher levels of pain.
Modified Morphine Equivalent (MME) differences | 7 days
  Total morphine milligram equivalents (MME) will be assessed
hospital-free days | 30 days
  number of outpatient days for 1 month following randomization
spirometry values | 7 days
  measurements of inspiratory volume in milliliters will be taken pre-placement, 60 minutes after catheter insertion, the following day, and each subsequent morning
mean respiratory rates | 7 days
  number of inspiratory cycles per minute taken each day until the patient is discharged
Patient reported quality of life | 7 days
  Patient reported quality of life will be measured through the EuroQol instrument (EQ-5D-5L). The EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "no problems" through "extreme problems."

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Warriner, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No